CLINICAL TRIAL: NCT06445088
Title: Evaluation of Diagnostic Performance of a Detection Kit for Epstein-Barr Virus C Promoter Methylation in Nasopharyngeal Carcinoma
Brief Title: Diagnostic Accuracy of EBV C Promoter Methylation Kit in Nasopharyngeal Carcinoma
Status: Recruiting | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Collaborators: Fujian Cancer Hospital (Other Government); Wuzhou Red Cross Hospital (Other); Zhongshan People's Hospital, Guangdong, China (Other); First Affiliated Hospital of Guangxi Medical University (Other)
Responsible Party: Principal Investigator, Hai-Qiang Mai,MD,PhD, Principal Investigator, Sun Yat-sen University
Other Study IDs: YKP2023-02-04
Record Dates: First submitted 2024-05-27; First posted 2024-06-06 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Nasopharyngeal Carcinoma; Diagnosis; Methylation Detection; Epstein-Barr virus
MeSH Terms: conditions — Nasopharyngeal Carcinoma; Disease; Epstein-Barr Virus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples With DNA — Blood and nasopharyngeal swabs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Diagnosis cohort: The participant has signs or symptoms suggestive of nasopharyngeal carcinoma, or has a condition that needs to be differentiated from nasopharyngeal carcinoma
  Interventions: Diagnostic Test: VCA-IgA, EBNA1-IgA, and EBV-DNA; Diagnostic Test: EBV C Promoter Methylation Detection in nasopharyngeal swab samples

INTERVENTIONS:
Diagnostic Test: VCA-IgA, EBNA1-IgA, and EBV-DNA — Detect VCA-IgA, EBNA1-IgA, and EBV-DNA for all participants.
Diagnostic Test: EBV C Promoter Methylation Detection in nasopharyngeal swab samples — Detection of methylation status of Epstein-Barr virus C promoter in human nasopharyngeal swab samples

SUMMARY:
This clinical study aims to evaluate the diagnostic performance of a new Epstein-Barr virus (EBV) C promoter methylation detection kit. All participants will undergo a series of diagnostic tests including VCA-IgA, EBNA1-IgA, and EBV-DNA assays. Additionally, nasopharyngeal swabs will be analyzed for EBV C promoter methylation. Confirmatory biopsy will be performed on all patients to establish a definitive diagnosis. This comprehensive approach seeks to assess the effectiveness of the methylation detection kit in a clinical setting.

ELIGIBILITY:
Inclusion Criteria:

Participants who meet the following Article 1 and also meet one of Articles 2 to 6 can be enrolled:

* Understand, sign, and date the informed consent document to participate in the study
* Display one or more symptoms or signs indicative of nasopharyngeal carcinoma
* Test positive for EBV antibodies or EBV DNA
* Be diagnosed with other head and neck carcinomas
* Be diagnosed with malignancies associated with EBV infection
* Require differential diagnosis from nasopharyngeal carcinoma during endoscopic or other imaging examinations
* Fulfill any additional conditions deemed appropriate by the investigator for inclusion in this study

Exclusion Criteria:

* Have been diagnosed with nasopharyngeal carcinoma and have undergone treatment
* Experience relapse or metastasis of nasopharyngeal carcinoma following treatment
* Have unsuccessful nasopharyngeal swab collections
* Present any other conditions considered by the investigator as unsuitable for participation in this trial

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population includes individuals suspected of having nasopharyngeal carcinoma or who may be confused with nasopharyngeal carcinoma cases.
Sampling Method: Non-Probability Sample
Enrollment: 908 (Estimated)
Dates: Start 2024-05-29 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of Epstein-Barr Virus C Promoter Methylation in Diagnosing Nasopharyngeal Carcinoma | From enrollment to final diagnosis, up to 4 weeks
  Measure the sensitivity of Epstein-Barr Virus (EBV) C Promoter Methylation as a diagnostic marker for Nasopharyngeal Carcinoma (NPC). Sensitivity will be calculated as the proportion of true positive cases (patients correctly identified with NPC) out of the total number of actual NPC cases.
Specificity of Epstein-Barr Virus C Promoter Methylation in Diagnosing Nasopharyngeal Carcinoma | From enrollment to final diagnosis, up to 4 weeks
  Measure the specificity of Epstein-Barr Virus (EBV) C Promoter Methylation as a diagnostic marker for Nasopharyngeal Carcinoma (NPC). Specificity will be calculated as the proportion of true negative cases (patients correctly identified without NPC) out of the total number of actual non-NPC cases.
Kappa Value of Epstein-Barr Virus C Promoter Methylation in Diagnosing Nasopharyngeal Carcinoma | From enrollment to final diagnosis, up to 4 weeks
  Evaluate the agreement between Epstein-Barr Virus (EBV) C Promoter Methylation and the gold standard diagnostic methods for Nasopharyngeal Carcinoma (NPC) using the Kappa statistic. The Kappa value will indicate the consistency and reliability of EBV C Promoter Methylation as a diagnostic tool compared to established diagnostic criteria.
Concordance Analysis of Test Reagents and Sequencing Methods in EBV C Promoter Methylation Detection | From enrollment to final diagnosis, up to 4 weeks
  This measure evaluates the positive, negative, and total concordance rates, as well as the Kappa Value, between test reagents and two established sequencing techniques-Sanger sequencing and pyrosequencing-for detecting Epstein-Barr virus C promoter methylation. The accuracy of these detection methods is assessed by comparing their results to those obtained through the widely used and mature technologies of Sanger dideoxy chain termination and pyrosequencing, often considered the "gold standards" for gene sequence analysis. This study aims to evaluate the reliability and accuracy of the test reagents in identifying methylation of the EBV C promoter, using these established sequencing benchmarks.

SECONDARY OUTCOMES:
Concordance Rates between EBV-Related Antibodies and EBV C Promoter Methylation | From enrollment to final diagnosis, up to 4 weeks
  This outcome measures the agreement rates between EBV C promoter methylation and EBV-related antibodies in the diagnosis of nasopharyngeal carcinoma without a gold standard for comparison. It includes an evaluation of the positive concordance rates, negative concordance rates, and Kappa value, which might reflect limited conclusiveness but offer insight into the relative alignment of these diagnostic tests. This will help ascertain their comparative reliability and diagnostic utility in a real-world setting.
Concordance Rates between EBV-DNA and EBV C Promoter Methylation | From enrollment to final diagnosis, up to 4 weeks
  This outcome measures the agreement rates between EBV C promoter methylation and EBV-DNA in the diagnosis of nasopharyngeal carcinoma without a gold standard for comparison. It includes an evaluation of the positive concordance rates, negative concordance rates, and Kappa value, which might reflect limited conclusiveness but offer insight into the relative alignment of these diagnostic tests. This will help ascertain their comparative reliability and diagnostic utility in a real-world setting.

OTHER OUTCOMES:
Dynamics of EBV C Promoter Methylation Before and After Nasopharyngeal Carcinoma Treatment | From enrollment to the end of treatment at 6 months, up to 1 years
  During follow-up consultations 1 to 6 months post-discharge, nasopharyngeal swabs will be collected to observe the dynamics of EBV C promoter methylation before and after treatment for nasopharyngeal carcinoma

CONTACTS AND LOCATIONS:
Overall Officials: Hai-Qiang Mai, Study Chair — Sun Yat-sen University; Zhen-Zhou Xiao, Principal Investigator — Fujian Cancer Hospital; Min-Zhong Tang, Principal Investigator — Wuzhou Red Cross Hospital; Min-Yi Fu, Principal Investigator — Zhongshan People's Hospital, Guangdong, China; Zhe Zhang, Principal Investigator — First Affiliated Hospital of Guangxi Medical University
Locations (5):
- China (5):
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong
  - ZhongShan City People's Hospital, Zhongshan, Guangdong
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - Wuzhou Red Cross Hospital, Wuzhou, Guangxi

IPD SHARING:
Plan to Share IPD: No